CLINICAL TRIAL: NCT01963689
Title: Aromatherapy for Anxiety and Self-esteem: Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Juliana Rizzo Gnatta, Juliana Rizzo Gnatta, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 469376
Record Dates: First submitted 2013-10-13; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Anxiety; Self Esteem
Keywords: Anxiety; Self-Esteem
MeSH Terms: conditions — Anxiety Disorders | interventions — Massage; Aromatherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention Group 2 (Placebo Comparator): Individuals belonging to Group 2 received a bottle containing aromatic gel enriched with ylang ylang essence only in 2% concentration and used massage with essential oil 3 times a day: leaving home to go to work, leaving the shift and before bedtime. The points indicated were the two handles and the sternum. Gel was applied and massaged in a circular motion for 30 seconds.
  Interventions: Other: Intervention Group 2
- Intervention Group 1 (Experimental): Individuals belonging to Group 1 received a bottle containing aromatic gel enriched with essential oil of ylang ylang in a concentration of 2% and used massage with essential oil 3 times a day: leaving home to go to work, leaving the shift and before bedtime. The points indicated were the two handles and the sternum. Gel was applied and massaged in a circular motion for 30 seconds.
  Interventions: Other: Intervention Group 1
- Intervention Group 3 (Experimental): The subjects in Group 3 were responsible for before the beginning of their working, put a drop of essential oil of ylang ylang in cotton located within the freshener personal and should be used throughout your work shift
  Interventions: Other: Intervention Group 3

INTERVENTIONS:
Other: Intervention Group 2 — Massage with Ylang Ylang Essence was applied for 30 seconds on the handle and the sternum area
  Other Names: Massage; Aromatherapy
  Arms: Intervention Group 2
Other: Intervention Group 1 — Massage with Ylang Ylang essential oil in the wrist and in the region of the sternum
  Other Names: Massage; Aromatherapy
  Arms: Intervention Group 1
Other: Intervention Group 3 — Put a drop of essential oil of ylang ylang in cotton located within the freshener and inhale throughout their work shift
  Other Names: Aromatherapy
  Arms: Intervention Group 3

SUMMARY:
The aim of this study was to determine whether the use of Ylang Ylang essential oil through dermal application or inhalation alters the perception of anxiety and self-esteem and physiological parameters such us blood pressure and temperature.

DETAILED DESCRIPTION:
34 nurses from the University Hospital participated in this study and were randomized into three groups: one that received the Ylang Ylang Essential Oil cutaneous route, the second received the Essential Oil inhalation and the third (placebo) received the essence of Ylang ylang cutaneous route.

ELIGIBILITY:
Inclusion Criteria:

* be an employee of the nursing team and not be on probation
* accept make use gel or freshener containing essential oil or essence ylang ylang
* respond Anxiety Inventory(STAI)and Self-esteem scale and present moderate, high or very high anxiety on the STAI, medium or low self-esteem on the scale Self-esteem
* accept not wear perfume during the survey period
* accept the smell of Ylang Ylang.

Exclusion Criteria:

* Self reported Hypotension
* Medical License or vacation during the period

Ages: 34 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | after 60 days
  The State-Trait Anxiety Inventory consists of 2 scales, each one containing 20 items. One of the scales evaluates state anxiety, characterized by subjective feelings of tension and apprehension, followed by autonomic nervous system responses at a given moment. Trait anxiety, assessed by the other scale, refers to a relatively stable tendency to perceive situations at threatening and react anxiously to them. The scores are divided into low, moderate, high and very high and are determined by the sum of 20 symptoms from a 5-point Likert-type scale.The range of scores is 20-80, the higher the score indicating greater anxiety for both the Trait and State Anxiety.

SECONDARY OUTCOMES:
Self-Esteem Scale | after 60 days
  This is a unidimensional measure of self-esteem, which has 15 statements about the assessments that the subject makes about itself. For each statement, the subject chooses one of two options: agree or disagree. The level of self-esteem is provided through a template that assigns one point for each answer in agreement and zero points for each answer in disagreement. The maximum score is 15 points and the minimum is 0 points.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Júlia P da Silva, Principal Investigator — Nursing School of São Paulo University